CLINICAL TRIAL: NCT00288470
Title: A Double-blinded Evaluation of Safety and Efficacy of Hylaform and Hylaform Plus Compared to Zyplast.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Purpose: Treatment
Other Study IDs: HYLA-001-01
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Facial Wrinkles

INTERVENTIONS:
Device: Hylaform, Hylaform Plus (hylan B gel)

SUMMARY:
A clinical study to investigate the safety and efficacy of Hylaform and Hylaform Plus for correction of facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* bilateral nasolabial folds with severity score 3 or 4 on the 6-point grading scale

Exclusion Criteria:

* pregnant/lactating women
* patients who previously received permanent facial implants or using ovet-the-counter products

Ages: 30 Years to 55 Years | Sex: All
Age Groups: Adult
Dates: Start 2002-06; Study Completion 2003-08

PRIMARY OUTCOMES:
Non-inferiority as compared to standard of care as assigned by blinded reviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company